CLINICAL TRIAL: NCT02349165
Title: Standard Versus Transepithelial Corneal Crosslinking for Treatment of Progressive Keratoconus
Brief Title: Standard Versus Transepithelial Corneal Crosslinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nienke Soeters (Other)
Collaborators: Dr. F.P. Fischer Stichting (Unknown); Stichting Nederlands Oogheelkundig Onderzoek (Unknown)
Responsible Party: Sponsor-Investigator, Nienke Soeters, BOptom, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL29961; 10-374 (Registry Identifier: METC UMC Utrecht)
Record Dates: First submitted 2015-01-17; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- epithelium off CXL (Active Comparator): epithelium removal + 30 minute isotonic riboflavin eye drops (3 minute interval) + 30 minutes ultraviolet-A irradiation (riboflavin every 5 minutes)
  Interventions: Procedure: Transepithelial versus epithelium-off CXL; Drug: Isotonic riboflavin
- Ricrolin TE CXL (Experimental): Ricrolin-TE eye drops for 15 minutes (2 minute interval) and 15 minute Ricrolin TE pooled on the cornea using a silicone ring + 30 minutes ultraviolet-A irradiation (Ricrolin TE every 5 minutes).
  Interventions: Procedure: Transepithelial versus epithelium-off CXL; Drug: Ricrolin TE

INTERVENTIONS:
Procedure: Transepithelial versus epithelium-off CXL — A comparison of the CXL procedure with and without epithelium removal
  Other Names: epithelium-on versus epithelium-ff corneal crosslinking
Drug: Ricrolin TE — Ricrolin TE was instilled during 30 minutes before ultraviolet-A irradiation
  Arms: Ricrolin TE CXL
Drug: Isotonic riboflavin — After epithelium removal, isotonic riboflavin was instilled during 30 minutes before ultraviolet-A irradiation
  Arms: epithelium off CXL

SUMMARY:
The gold standard corneal crosslinking (CXL) technique involves the initial step of epithelial removal, in order to achieve a sufficient treatment effect (meaning: stabilisation of progressive keratoconus (KC). Our aim is to evaluate the effects of transepithelial CXL (TE-CXL), whereby the epithelium is left intact and the cornea is instead treated by a solution composed of 0.1% riboflavin, combined with enhancers, after which standard CXL is performed. This solution seems to facilitate riboflavin penetration into the corneal stroma through the intact epithelium. The investigators expect to achieve a similar effect of TE-CXL with the advantage of a faster healing time and less risk of infections.

ELIGIBILITY:
Inclusion Criteria:

* Documented progressive KC (by Pentacam and/or corneal topography imaging).
* A clear central cornea.
* A minimal corneal thickness of ≥ 400 µm at the thinnest corneal location (Pentacam imaging).
* Minimal Snellen corrected distance visual acuity of ≥ 0.4.
* Patient age of ≥ 18 years.

For this research study, the inclusion parameters will be the same as mentioned above, with the following additional inclusion criteria:

* Documented progression of KC, as demonstrated by anterior segment imaging and/or corneal topography:

  o Defined an increase in maximal keratometry, steepest keratometry, mean keratometry or topographic cylinder value by ≥ 0.5 D over the previous 6 months and/or a decrease in thinnest pachymetry
* Documented progression of KC defined by increase in refractive cylinder of ≥ 0.5 D over the previous 6 months

Exclusion Criteria:

* Presence of corneal scars.
* History of epithelial healing problems.
* Presence of previous ocular infection (such as herpes keratitis).
* Patients who are pregnant and/or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Clinical stabilisation of keratoconus one year after CXL | 1 year
  Using a Scheimpflug device (Pentacam, Oculus), topography measurements are performed. Clinical stabilisation is defined as an increase of no more than 1 diopter of the maximum keratometry value over the preoperative maximum keratometry value.

SECONDARY OUTCOMES:
Complications, defined as epithelial healing problems and/or keratitis. | 1 year
  the incidence of epithelial healing problems after treatment will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558